CLINICAL TRIAL: NCT04145128
Title: A Phase 1, Open-Label, Single Ascending Dose Study to Evaluate AG-881 in Healthy Japanese and Non-Asian Subjects
Brief Title: A Study to Evaluate AG-881 in Healthy Japanese and Non-Asian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AG881-C-008
Record Dates: First submitted 2019-10-29; First posted 2019-10-30 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetic study; AG-881
MeSH Terms: interventions — vorasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AG-881 (Experimental): Participants will receive AG-881 10 mg, tablet orally, once in Period 1 followed by AG-881 50 mg, tablet orally, once in Period 2. Period 1 and Period 2 will be separated by a washout period of 20 days between doses.
  Interventions: Drug: AG881

INTERVENTIONS:
Drug: AG881 — AG-881 tablets.
  Other Names: Vorasidenib; AGI 23088; AGI 0023088

SUMMARY:
The purpose of this study is to compare the pharmacokinetics (PK) and safety of AG-881 in healthy Japanese and Non-Asian participants after single oral doses of 10 mg and 50 mg of AG-881.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided voluntary written informed consent.
2. Adult male or female, 18 to 55 years of age, inclusive, at Screening.
3. Continuous nonsmoker who has not used nicotine containing products for at least 3 months prior to the first dosing and throughout the study.
4. Have a body mass index (BMI) of ≥ 18.0 and ≤ 32.0 kg/m^2 at Screening.
5. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECG. Liver function tests (serum alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase [ALP], and bilirubin [total and direct]) must be ≤ the upper limit of normal (ULN).
6. Female participants must be of nonchildbearing potential defined as a female who has undergone one of the following sterilization procedures at least 6 months prior to the first dosing: hysteroscopic sterilization; bilateral tubal ligation or bilateral salpingectomy; hysterectomy; bilateral oophorectomy. Or is postmenopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
7. A nonvasectomized, male participant must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing of study drug. A male who has been vasectomized less than 4 months prior to study first dosing must follow the same restrictions as a nonvasectomized male).
8. Male participants must agree not to donate sperm from the first dosing until 90 days after the last dosing.
9. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.
10. Additional Criteria for Japanese participants only: be first-generation Japanese, defined as meeting all of the following conditions: born in Japan; has 2 Japanese biological parents and 4 Japanese biological grandparents; has lived outside of Japan for <5 years; has made no significant changes in lifestyle, including diet, since leaving Japan.
11. Additional Criteria for Non-Asian participants only: Non-Asian participants will have 2 biological parents and 4 biological grandparents of Non-Asian descent.

Exclusion Criteria:

1. Mentally or legally incapacitated or has significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. History of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or pose an additional risk to the participant (eg, history or presence of rashes) by their participation in the study.
4. History of stomach or intestinal surgery that would potentially alter absorption/secretion; or any major surgical procedure within the previous 3 months prior to Screening.
5. History of severe and/or uncontrolled ventricular arrhythmias, or other factors that increase the risk of QT prolongation or arrhythmic events (eg, heart failure, hypokalemia, family history of long QT interval syndrome).
6. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
7. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
8. Any positive responses on the Columbia-Suicide Severity Rating Scale (C-SSRS).
9. Female participants of childbearing potential.
10. Female participants with a positive pregnancy test or who are lactating.
11. Positive urine drug or alcohol results at Screening or Day -1/Day 21.
12. Positive results at Screening for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV) antibodies.
13. QTcF interval is >450 msec, or QRS interval >110 msec, or PR interval >220 msec, or participants who have ECG findings deemed abnormal with clinical significance by the Investigator or designee at Screening.
14. Supine blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at Screening.
15. Supine heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at Screening.
16. Estimated creatinine clearance <90 mL/min at Screening.
17. Unable to refrain from or anticipates the use of: any drug, including prescription and non-prescription medications, herbal remedies, and vitamin supplements, beginning 14 days prior to the first dosing and throughout the study. After first dosing, acetaminophen (<2 g per 24 hour) may be administered at the discretion of Investigator or designee. Hormone replacement therapy will not be allowed; any drugs known to be strong inducers of CYP3A, CYP2C9, or CYP2C19 enzymes including St. John's Wort and/or, gastric acid reducing agents (eg, protonpump inhibitors, H2-receptor antagonists, antacids) for 28 days, or drugs that can prolong the QT interval for 28 days, prior to the first dosing and throughout the study. Appropriate sources (eg, Flockhart TableTM) will be consulted to confirm lack of PK/Pharmacodynamic (PD) interaction with study drug.
18. Refuses to abstain from alcohol from 48 hours prior to the first dosing and throughout the study.
19. Refuses to abstain from grapefruit-containing foods or beverages or Seville orange containing foods or beverages from 14 days prior to the first dosing and throughout the study.
20. Donation of blood or significant blood loss within 56 days prior to the first dose.
21. Plasma donation within 7 days prior to the first dose.
22. Receipt of blood or blood products within 2 months prior to the first dose.
23. Participation in another clinical study within 30 days prior to the first dose. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve from Time Zero to the Time of the Last Measurable Concentration (AUC0-last) of AG881 | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-∞) of AG881 | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Clearance Following Extravascular Dosing (CL/F) of AG881 | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Maximum Plasma Concentration Observed (Cmax) of AG881 | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Terminal Elimination Half-life (t1/2) of AG881 | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Time of Maximum Plasma Concentration (tmax) of AG881 | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881
Apparent Volume of Distribution (Vd/F) of AG881 | Pre-dose and multiple time points post-dose (up to 504 hours) after each administration of AG-881

SECONDARY OUTCOMES:
Number of Participants with Changes in Clinical Laboratory Tests from Screening to 22 days in Period 1 and 2 | Screening (Day -1) up to 22 days in Period 1 and 2 (Each Period is 22 days)
  Clinical laboratory assessments will include hematology, blood chemistry, and urinalysis.
Number of Participants with Changes in Physical Examinations from Screening to 22 days in Period 1 and 2 | Screening (Day -1) up to 22 days in Period 1 and 2 (Each Period is 22 days)
  Physical examination will include, examination of skin, neurological, respiratory, cardiovascular, and gastrointestinal systems.
Number of Participants with Changes in Vital Sign Measurements from Screening to 22 days in Period 1 and 2 | Screening (Day -1) up to 22 days in Period 1 and 2 (Each Period is 22 days)
  Vital sign measurements will include body temperature, respiratory rate, blood pressure, and heart rate.
Number of Participants with Changes in Electrocardiograms (ECGs) from Screening to 22 days in Period 1 and 2 | Screening (Day -1) up to 22 days in Period 1 and 2 (Each Period is 22 days)
Number of Participants with Adverse Events (AEs) | Up to 28 days after last dose of AG-881 (Up to 71 days)
  An AE is any untoward medical occurrence associated with the use of a drug, whether or not considered drug-related.
Number of Participants Using Concomitant Medications | Up to 28 days after last dose of AG-881 (Up to 71 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- WCCT GLobal, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No